CLINICAL TRIAL: NCT06805890
Title: Study of Tissue Repair in Inflammatory Bowel Disease Exploiting Organoid Technology
Acronym: ORGANOIDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM24_0062; 2024-A00510-47 (Other: EUdraCT)
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases (IBD); Ulcerative Colitis (Disorder)
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): Patients of either sex aged 18 years or older and undergoing a screening colonoscopy in the context of a family history of colonic neoplasia, follow-up of colonic polyps or functional intestinal disorders OR undergoing intestinal resection for intestinal neoplasia, occlusive syndrome or colostomy
  Interventions: Procedure: Colonoscopy - biopsies in healthy tissue; Procedure: Surgical resection - healthy mucous membrane
- IBD group (Experimental): Patients of either sex aged 18 years or older with Crohn's Disease or ulcerative colitis in accordance with accepted clinical, endoscopic, histological and/or radiologic criteria, regardless of the level, severity of the disease or duration of disease progression or patients undergoing a screening colonoscopy in the context of IBD disease follow-up OR undergoing intestinal resection for IBD disease aggravation
  Interventions: Procedure: Colonoscopy - IBD inflamed tissue; Procedure: Surgical resection - IBD inflamed mucous membrane; Procedure: Surgical resection - healthy mucous membrane

INTERVENTIONS:
Procedure: Colonoscopy - IBD inflamed tissue — Collection of 10 colonic biopsies in IBD inflamed tissue
  Arms: IBD group
Procedure: Surgical resection - IBD inflamed mucous membrane — Collection of a portion of IBD inflamed mucous membrane
  Arms: IBD group
Procedure: Colonoscopy - biopsies in healthy tissue — Collection of 10 colonic biopsies in healthy tissue
  Arms: Control group
Procedure: Surgical resection - healthy mucous membrane — Collection of a portion of healthy mucous membrane

SUMMARY:
Inflammatory Bowel Diseases (IBD) are chronic inflammations of the gastrointestinal tract. Regardless of the etiology, a common trait of IBD pathogenesis is the inflammatory damage inflicted on the intestinal mucosa and the loss of intestinal epithelial barrier integrity. Therefore, understanding the mechanisms that govern IEC's capacity to maintain barrier function and to orchestrate mucosal healing is considered a major goal in translational research. The investigators are interested in understanding how the inflammatory environment present in the intestinal mucosa, of IBD patients influences epithelial cells capacity to govern repair. The complexities of the cytokine and metabolic milieu present in IBD patients render the study of the contribution of each cytokine, metabolite, and intracellular pathway extremely complicated. Therefore, most of the processes that govern tissue regeneration are studied with the use of mouse models that recapitulate one or multiple features of IBD and allow for genetical modifications of the gene and pathway of interest. While mouse models are uniquely suited to study the complex crosstalk between the immune system, the microbiota, and the intestinal epithelia, they introduce the important problem of species-specific differences, which can hamper the translational value of mouse studies.

To overcome these shortcomings, the investigators propose to explore the influence of cytokines and metabolites in digestive organoids derived from patients and controls. Importantly, it was demonstrated that gene expression and innate immune responses are altered in primary organoids derived from patients with IBD, including altered ability to proliferate, respond to cytokines, metabolic capacity, and efficiently form organoids suggesting that major differences between patient's and control's epithelial cell biology can be faithfully replicated in this system.

Given these premises, the investigators propose the following objectives:

Primary objective:

The main objective of this study is to establish that patient's epithelial cells from inflamed mucosae have decreased ability to repair the intestinal mucosa, as compared to epithelial cells from non-inflamed regions in the same patient, or to control subject with no inflammatory digestive diseases.

The investigators will explore this question both deriving organoids from clinical samples and exposing them to pro inflammatory cytokines and metabolites in vitro, as well as by analyzing repair responses from the aforementioned clinical samples ex vivo.

Secondary objective

The secondary goals of this study are:

- To compare organoids derived from: epithelia in inflamed mucosa of IBD patients, epithelia in non-inflamed mucosa of IBD patients, and epithelia from the mucosa of non-IBD controls in their capacity to mount a repair response in response to inflammatory cytokines or luminal metabolites.

Namely the investigators will evaluate the following parameters:

* Their capacity to proliferate.
* Their ability to survive treatment with pro-inflammatory cytokines
* The activation of intracellular pathways associated with cell death.
* Their overall metabolic activity.
* The balance between stem and differentiated epithelial cell types.
* The transcriptional activation of protective pathways such as those associated with proliferation, migration, differentiation and cell survival.
* To evaluate hallmarks of tissue repair in biopsies derived from epithelia in inflamed mucosa of IBD patients, epithelia in non-inflamed mucosa of IBD patients, and epithelia from the mucosa of non-IBD controls, and to correlate them to the levels of inflammatory cytokines, luminal metabolites and overall disease severity. Namely the investigators will evaluate the following parameters:
* The abundance of proliferating cells.
* The activation of intracellular pathways associated with cell death and survival.
* Their overall metabolic activity.
* The balance between stem and differentiated epithelial cell types.
* The transcriptional activation of protective pathways such as those associated with proliferation, migration, differentiation and cell survival.

ELIGIBILITY:
For IBD group the inclusion criteria will be:

* Patients of either sex aged 18 years or older
* Patient that have read the information form and signed consent
* Patient covered with health insurance
* Patients with Crohn's Disease or ulcerative colitis in accordance with accepted clinical, endoscopic, histological and/or radiologic criteria, regardless of the level, severity of the disease or duration of disease progression.
* Patients with colonic involvement of Crohn's disease or ulcerative colitis
* Patients undergoing a screening colonoscopy in the context of IBD disease follow-up OR undergoing intestinal resection for IBD disease aggravation

For control group the inclusion criteria will be:

* Patients of either sex aged 18 years or older
* Patient that have read the information form and signed consent
* Patient covered with health insurance
* Patients undergoing a screening colonoscopy in the context of a family history of colonic neoplasia, follow-up of colonic polyps or functional intestinal disorders OR undergoing intestinal resection for intestinal neoplasia, occlusive syndrome or colostomy

The non-inclusion criteria for IBD group will be:

* Contraindication to the anaesthetic or colonoscopy procedure
* Patients without colonic involvement of Crohn's disease or ulcerative colitis
* Patients of Adults without legal capacity
* Patients in Health and Social Establishments
* Persons in emergency situations
* Persons deprived of their liberty
* Non-affiliated to a social security scheme
* Absence or refusal of the informed consent

The non-inclusion criteria for control group will be:

* IBD disease revealed during colonoscopy or gastrointestinal resection
* Patient suffering from Immune-Mediated Inflammatory Diseases (IMIDs)
* Contraindication to the anaesthetic or colonoscopy procedure
* Patients of Adults without legal capacity
* Patients in Health and Social Establishments
* Persons in emergency situations
* Persons deprived of their liberty
* Non-affiliated to a social security scheme
* Absence or refusal of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-03-24 (Estimated); Study Completion 2027-03-24 (Estimated)

PRIMARY OUTCOMES:
Repair status of IBD patient's epithelial cells from inflamed mucosae | From enrollmet to the end of following at 1 month
  To establish that patient's epithelial cells from inflamed mucosae have decreased ability to repair the intestinal mucosa, as compared to epithelial cells from non-inflamed regions in the same patient, or to control subject with no inflammatory digestive diseases

SECONDARY OUTCOMES:
Evaluate the molecular mechanism involved in the reduced capacity of epithelial cells of IBD patients to repair intestinal mucosa | From enrollment to the end of following at 1 month
  Evaluation of:
  * The capacity epithelial cells of IBD patients to proliferate: ratio of Ki67+cells.
  * The ability of epithelial cells of IBD patients to survive treatment with pro-inflammatory cytokines: ratio between live and dead organoids.
  * The activation of intracellular pathways associated with cell death: relative quantification of biochemical activation of 1) apoptotic caspases,2) pyroptosis effectors (GSDMs),3) Necroptosis effectors (MLKL).
  * The balance between stem and differentiated epithelial cell types: the relative gene expression of the stemness associated genes LGR5, OLFM4, and the hallmark genes of differentiated cell types AQP8, MUC2, LYZ1, CHGA).
Genetically determine the involvement of cell death and protective pathways that reduce repair capacity in patients. | From enrollment to the end of following at 1 month
  After a genetically modify with CRISPR-CAS9 technology:
  * The capacity of modified epithelial cells of IBD patients to proliferate: ratio of Ki67+cells.
  * The ability of modified epithelial cells of IBD patients to survive treatment with pro-inflammatory cytokines: ratio between live and dead organoids.
  * The activation of intracellular pathways associated with cell death: relative quantification of biochemical activation of 1) apoptotic caspases,2) pyroptosis effectors (GSDMs),3) Necroptosis effectors (MLKL).
  * The balance between stem and differentiated epithelial cell types: the relative gene expression of the stemness associated genes LGR5, OLFM4, and the hallmark genes of differentiated cell types AQP8, MUC2, LYZ1, CHGA).
3. Explore the activation of molecular mechanisms identified in patient biopsies and correlate them with the inflammatory environment present in the patient's tissues | From enrollment to the end of following at 1 month
  * Proliferation in FFPE biopsies and RNA from RNAlater fixed biopsies: Ki67 upregulation by immunohistochemistry (IHC), PCNA gene expression, Proliferation transcriptional signature by RNAseq etc…).
  * Cell death by biochemical analysis of cell death pathways by Western Blot (WB) and IHC in flash frozen biopsies: relative quantification of biochemical activation of 1) apoptotic caspases; 2) pyroptosis effectors (GSDMs); 3) Necroptosis effectors (MLKL).
  * Differentiation status of epithelial cells from DMSO conserved biopsies: staining of cell type markers by IHC, scRNAseq of dissociated epithelial cells.
  * The metabolic landscape of epithelial cells in flash frozen biopsies: the metabolome of the cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Nord Hospital, Marseille, France

IPD SHARING:
Plan to Share IPD: No